CLINICAL TRIAL: NCT05972590
Title: Interventional, With Minimal Risks and Constraints Study Aiming at Constituting a Biological Samples Collection Constituted From Volunteers Aged Between 50 and 75 Years Old And Used For Scientific Purposes
Brief Title: Characterization of Fecal Microbiota in a Population Aged 50 to 75 Years Targeted by Seasonal Vaccination
Acronym: FIFTY+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioaster (Other)
Collaborators: BioFortis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-A00947-38
Record Dates: First submitted 2023-07-10; First posted 2023-08-02 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Elderly Volunteers
Keywords: Biobank; Health Ageing; Blood, TruCultures; Stools; Strain isolation; Probiotics; Immunity; Vaccination
MeSH Terms: interventions — Blood Specimen Collection; Defecation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 50-75 years old volunteers cohort (Other): Biological samples collection Blood drawing + faeces collection
  Interventions: Other: Biological samples collection (blood + feces)

INTERVENTIONS:
Other: Biological samples collection (blood + feces) — Blood + stools samples will be collected from each volunteer

SUMMARY:
The goal of this interventional study is to constitute a biological samples collection collected from healthy elderly volunteers and used for scientific purposes.

The main questions it aims to answer are:

* Improving knowledge of the composition of the gut microbiota
* Identify, isolate and culture microbiota species of interest in the field of health ageing or used as therapeutics associated to the vaccination
* Determining the correlation between the gut microbiota composition and the immune response of individuals.

DETAILED DESCRIPTION:
The compositional analysis of commensal bacterial populations collected from a variety of clinical samples has been recently made possible with the availability of Next Generation Sequencing (NGS) technologies. The term 'next-generation probiotics' (NGP) is now widely used to describe these commensal species of potential health interest.

However, this approach is still hampered by the fact that there are usually few or even no strains available for a number of commensal species.

In this context, BIOASTER has developed a specific technological process based on flow cytometry analysis and then sorting under strictly anaerobic conditions to target and cultivate commensal species of interest.

The goal of this study is to constitute a biological samples collection from elderly people, to proceed with the isolation of beneficial commensal strains such as Faecalibacterium prausnitzii, Akkermansia muciniphila and Oscillospiraceae, in a non-limitative way.

BIOASTER's objective is to strengthen technological support, provide new knowledges and tools for the development of next-generation products. Numerous biotherapeutics companies will benefit from this pipeline, ultimately improving the chances of survival in life-threatening diseases with unmet medical needs.

Elderly people will be recruited by the investigational unit Biofortis.

Blood (Whole blood + TruCulture tubes) and feces will be collected from each volunteer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 50 and 75,
* BMI between 18.5 and 29 kg/m2,
* Normal clinical examination,
* Written consent obtained

Exclusion Criteria:

* Diagnosed acute or chronic gastrointestinal disease or complication (e.g., celiac disease, gastroesophageal reflux, gastric or duodenal ulcer, Crohn's disease, hemorrhoids, irritable bowel syndrome)
* Infectious gastrointestinal event within 3 months prior to inclusion
* Severe chronic disease (active cancer, HIV, severe renal failure, ongoing severe heart or liver or biliary disorders, arthritis) or severe chronic disease deemed incompatible with the conduct of the study by the investigator
* Major surgical procedure likely to disrupt the intestinal microbiota, within 6 months prior to inclusion
* Recent food allergy < 3 months prior to inclusion
* Antibiotic, antiviral, antifungal, proton pump inhibitor or any other treatment likely to disrupt the microbiota in the 3 months prior to inclusion
* Previous or current use of a treatment that may disrupt the microbiota (e.g. laxatives, antidiarrheals, antacids...) in the last 3 months
* Significant change in dietary habits or physical activities in the 3 months prior to inclusion
* Consumption of more than 2 standard glasses of alcoholic beverages per day
* Smoking > 20 cigarettes per day, illicit drug use,
* Daily use of non-steroidal anti-inflammatory drugs (NSAIDs)
* Severe psychiatric or neurological pathology
* Subject with liquid stools (Bristol Score = 7) or very hard stools (Bristol Score = 1)
* Any vaccination in the last month before inclusion
* Subject unable to understand the purpose of the research, answer questions and give their decision to participate in the study
* Subject already included in another research study involving the human subject
* Subject under guardianship and whose guardianship objects to the participation of his/her protectee,
* Subject not affiliated with a social security plan or not a beneficiary of such a plan

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Number and ratio of participants with per protocol collection of blood and feces | Baseline
  Number of volunteers included in the study and number blood/feces pairs collected.
Total number of bacteria strains collected | Baseline
  Isolation and culture of bacteria of interest in anaerobic conditions: constitution of a biobank of Akkermansia muciniphila, Faecalibacterium prausnitzii and Oscillospiraceae) for research purposes.
Fecal microbiome richness as assessed by alpha diversity | Baseline
  Genus and species of bacteria contained in the intestinal microbiota (alpha diversity calculation)

SECONDARY OUTCOMES:
Immunophenotyping of volunteers as assessed by cytokines quantification | Baseline
  serum samples will be analyzed by ELISA method to quantify cytokines
Immunophenotyping of volunteers as assessed by flow cytometry on immune cells | Baseline
  peripheral blood mononuclear cells will be stained with specific markers antibodies to characterize immune cells populations

CONTACTS AND LOCATIONS:
Overall Officials: Cyril GUYARD, Study Director — Bioaster; Stéphanie CAVIGIOLI, Principal Investigator — BioFortis
Locations (1):
- Biofortis, Paris, France

IPD SHARING:
Plan to Share IPD: No